CLINICAL TRIAL: NCT01084915
Title: The Results and Outcomes of the SAGB-VC in a High Volume Bariatric Centre
Brief Title: The Results and Outcomes of the Modified Swedish Adjustable Gastric Band (SAGB-VC)
Acronym: ROS
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Jens Homan, MD, Rijnstate Hospital
Other Study IDs: 680-070110-Aarts
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Weight Loss
Keywords: Weight loss after SAGB VC band placement
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SAGB VC group: Retrospectively patients with a SAGB-VC gastric band are inventorized. They will also be interviewed and BAROS scores will be taken.

SUMMARY:
Since a few years the SAGB-VC is used in our clinic. This type of band has a number of advantages when compared to the earlier versions of the adjustable gastric band (AGB), reducing the chances on leakage, tube disconnection and port problems. In our clinic the follow up is strict. All patients are required to follow a special follow-up program in which the patient is seen 19 times during the first two years after SAGB-VC placement.

This is the first retrospective clinical study of a large study population of >800 patients in which a SAGB-VC was placed. This study was conducted to evaluate the results and the efficiency of the SAGB-VC in our clinic.

ELIGIBILITY:
Inclusion Criteria:

* SAGB band placed from 2004-2008

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a SAGB-VC band from 2004-2008
Sampling Method: Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Weight loss | 2 months
  The amount of weight loss over time is researched

SECONDARY OUTCOMES:
Bariatric Analysis and Reporting Outcome System (BAROS) score | 2 months
  A specific score for quality of life (QOL) and outcome for bariatric surgery is inventorized
Operating time | 2 months
  Operating time is inventorized
Complications | 2 months
  Complications are inventorized
Co-morbidities | 2 months
  The reduction of co-morbidities is inventorized

CONTACTS AND LOCATIONS:
Overall Officials: F.J. Berends, MD, PhD, Principal Investigator — Rijnstate Hospital The Netherlands
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands